CLINICAL TRIAL: NCT07368569
Title: Investigation of the Effect of BI 764198 on the Pharmacokinetics of Metformin Following Multiple Oral Administration in Healthy Male and Female Trial Participants (an Open-label, Randomised, Two-way Crossover Trial)
Brief Title: A Study in Healthy People to Test Whether BI 764198 Influences the Amount of Metformin in the Body
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1434-0005; 2025-522432-14 (Registry Identifier: CTIS); U1111-1322-9764 (Registry Identifier: WHO Registry)
Record Dates: First submitted 2026-01-20; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Healthy
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference - Treatment (R-T) (Experimental): This arm starts with the reference treatment (R), metformin hydrochloride, followed by a washout period, and then the test treatment (T), metformin hydrochloride and BI 764198.
  Interventions: Drug: Metformin hydrochloride; Drug: BI 764198
- Treatment - Reference (T-R) (Experimental): This arm starts with the test treatment (T), metformin hydrochloride and BI 764198, followed by a washout period, and then the reference treatment (R), metformin hydrochloride.
  Interventions: Drug: Metformin hydrochloride; Drug: BI 764198

INTERVENTIONS:
Drug: Metformin hydrochloride — Metformin hydrochloride
Drug: BI 764198 — BI 764198

SUMMARY:
The main objective of this trial is to investigate the effect on the exposure of metformin in plasma when administered as an oral multiple dose together with multiple oral doses of BI 764198 (Test, T) as compared to when metformin is administered as an oral multiple dose alone (Reference, R).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female trial participant according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure [BP], Pulse rate [PR]), 12-lead Electrocardiogram (ECG), and clinical laboratory tests.
* Age of 18 to 55 years (inclusive).
* BMI of 18.5 to 29.9 kg / m² (inclusive).
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.
* Further inclusion criteria apply.

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator.
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 millimeters of mercury (mmHg), or pulse rate outside the range of 50 to 90 beat per minute (bpm).
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance.
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator.
* Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-03-17 (Estimated)

PRIMARY OUTCOMES:
Metformin: Area under the concentration-time (AUC) curve of the analyte in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) | Up to 5 days
Metformin: Maximum measured concentration of the analyte in plasma at steady state (Cmax,ss) | Up to 5 days

SECONDARY OUTCOMES:
Metformin: Renal clearance of the analyte from plasma at steady state (CL R,ss) | Up to 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com